CLINICAL TRIAL: NCT04105803
Title: Cardiac Mitochondrial Function After Heart Transplantation
Acronym: ENERGY-HTX
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Aarhus (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: 1-10-72-367-18
Record Dates: First submitted 2019-03-12; First posted 2019-09-26 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-07

CONDITIONS: Cardiac Allograft Vasculopathy; Acute Cellular Graft Rejection; Primary Graft Failure; Mitochondrial Function

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and endomyocardial biopsies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- De novo HTx: Procedure: Two perprocedural biopsies under transplantation is performed from the left ventricular septum.
  Procedure: Endomyocardial biopsies from the right ventricular septum, taken at scheduled standard HTx follow-up visits at our department (protocol is to take 4-5 biopsies, two additional biopsies will be taken at this visit).
  Procedure: is part of the scheduled standard HTx follow-up visits. This recording will be used for CAV evaluation. In addition to the protocol procedure, we will evaluate the hemodynamic status in the patients.
  Diagnostic test: Echocardiography and coronary angiography is part of the scheduled standard HTx follow-up visits.
- Longterm HTx: Procedure: Endomyocardial biopsies from the right ventricular septum, taken at scheduled standard HTx follow-up visits at our department (protocol is to take 4-5 biopsies, two additional biopsies will be taken at this visit).
  Procedure: Coronary Angiography is part of the scheduled standard HTx follow-up visits. This recording will be used for CAV evaluation. In addition to the protocol procedure, we will evaluate the hemodynamic status in the patients.
  Diagnostic test: Echocardiography is part of the scheduled standard HTx follow-up visits. No additional examinations will be performed. We will use the standard recordings to calculate the desired parameters.
- PET-scan de novo HTx: Radiation: Two PET-scans with 11C-acetate tracer will be performed.
  Procedure: Two perprocedural biopsies under transplantation is performed from the left ventricular septum.
  Procedure: Endomyocardial biopsies from the right ventricular septum, taken at scheduled standard HTx follow-up visits at our department (protocol is to take 4-5 biopsies, two additional biopsies will be taken at this visit).
  Procedure: Coronary Angiography is part of the scheduled standard HTx follow-up visits. This recording will be used for CAV evaluation. In addition to the protocol procedure, we will evaluate the hemodynamic status in the patients.
  Diagnostic test: Echocardiography is part of the scheduled standard HTx follow-up visits. No additional examinations will be performed. We will use the standard recordings to calculate the desired parameters.

SUMMARY:
Studies have shown that cardiac function is affected immediately after heart transplantation (HTx), but seems to recover to some extent over the first year. This immediate effect is associated with lack of oxygen in the tissue and reperfusion injury causing cellular energy depletion, mitochondrial failure and cellular damage. This condition may progress into full blown primary graft failure (PGF), characterized as deterioration of the transplanted heart, which is seen in 3-30 % of HTx patients. In addition to PGF, chronic rejection owing to cardiac allograft vasculopathy (CAV) may develop.

PGF and CAV remain the major heart related mortality causes, and additional assessment and treatments are therefore needed.

Acute cellular rejection (ACR) is diagnosed based on endomyocardial biopsies (EMB), which are routinely performed to ensure prober immunosuppression in HTx patients. ACR occur in approximately 25% of HTx patients, and is associated with PGF and CAV. However, mitochondrial function and integrity may prove to be a more sensitive marker of allograft rejection than endomyocardial biopsies. Therefore, assessment of mitochondrial function may allow for earlier detection of allograft rejection and dysfunction. This may be of particular importance as emerging treatments are targeting both energy substrate supply for adenosine-triphosphate generation produced by the mitochondria and mitochondrial function in the failing heart.

Despite the association between graft rejection and mitochondrial function, it remains unsettled whether mitochondrial function associate with PGF, ACR and CAV. Such findings may be of prognostic importance and even elucidate new treatment targets. Hence, we evaluate the mitochondrial status in HTx patients through four studies designed to assess different aspects of the interplay between cardiac function and mitochondrial integrity and function.

Hypotheses:

Study 1: Primary graft pump function is correlated to mitochondrial function in the first myocardial biopsy taken from the donor heart during the operation.

Study 2: Cardiac mitochondrial function improves over the first 3 months after a heart transplantation.

Study 3: Heart transplant patients with moderate to severe coronary graft vasculopathy has impaired mitochondrial function.

Study 4: Myocardial external energy efficiency by positron-emission tomography can be used as a marker of mitochondrial function and chronic rejection in HTx patients.

DETAILED DESCRIPTION:
Background

The prognosis after heart transplantation (HTx) has improved considerably since the first HTx was performed in 1967. Studies from our group have shown both left and right ventricular function is affected immediately after heart transplantation, but this seems to recover to some extent over the first year. This immediate effect on the graft organ following HTx is associated with tissue ischemia and reperfusion injury causing cellular energy depletion, mitochondrial failure and subsequent apoptosis. The condition may progress into full blown primary graft failure (PGF) with a need for mechanical cardiovascular support or inotropes which is seen in 3-30 % of HTx patients. The cardiac injury will consequently increase the risk of morbidity as well as mortality. In addition to acute PGF, a chronic rejection owing to coronary arterial vasculopathy (CAV) may develop. Hence, despite advances in peritransplantation treatment and immunosuppression, PGF and CAV remain the major heart related mortality causes following HTx and additional assessment and treatments are therefore needed.

Graft rejection is diagnosed, and the severity graded based on endomyocardial biopsies (EMB) taken percutaneously through the jugular or femoral veins. These biopsies are routinely performed at our institution to ensure prober immunosuppression following HTx.1 Acute cellular rejection (ACR) may occur in approximately 25% of the patients which is associated with PGF, CAV and later chronic rejection. However, mitochondrial function and integrity may prove to be a more sensitive marker of allograft rejection. In heart failure, mitochondria density changes while function and integrity is impaired linking the failing heart to energy deprivation. Animal studies demonstrate that deterioration in total mitochondrial function precedes histopathological changes during cardiac graft rejection following HTx. Therefore, assessment of mitochondrial function following HTx may allow for earlier detection of rejection and allograft dysfunction. This may be of particular importance as emerging treatments are targeting both energy substrate supply for adenosine-triphosphate (ATP) generation produced by the mitochondria as well as mitochondrial function in the failing heart. At our institution, we have established methods to evaluate mitochondrial function in myocardial tissue, and pilot studies have demonstrated feasibility with the use of EMB. In addition, by use of non-invasive 11C-acetate positron-emission tomography (PET), we can assess myocardial external energy efficiency (MEE) calculated by the ratio of myocardial external work (EW) and oxidative metabolism (MVO2). Thus, enabling quantification of coupling between mitochondrial energy production and mechanical work.

Despite the overt association between graft dysfunction/rejection and mitochondrial function, it remains unsettled whether mitochondrial content and function associate with PGF, ACR and CAV. Such findings may be of prognostic importance and even elucidate a new treatment target.

Hypotheses

1. Primary graft pump function is correlated to mitochondrial function in the first myocardial biopsy taken from the donor heart during the operation
2. Cardiac mitochondrial function improves over the first 3 months after a heart transplantation
3. Heart transplant patients with moderate to severe coronary graft vasculopathy has impaired mitochondrial function
4. MEE can be used as a marker of mitochondrial function and chronic rejection in HTx patients

Objectives

Study 1: To examine whether primary myocardial function is related to cardiac mitochondrial function in de novo HTx patients

Study 2: To investigate whether cardiac mitochondrial function improves over time after HTx along with improvement of cardiac function

Study 3: To examine whether heart transplanted patients with chronic rejection and graft vasculopathy have impaired mitochondrial function

Study 4: To evaluate whether MEE can be used as marker of mitochondrial function and chronic rejection

Design and endpoints

Study 1: The association between cardiac and mitochondrial function following HTx

Design: Myocardial mitochondrial function analyzed from 15 HTx patients taken from the donor heart during the transplantation will be compared to EMB from 15 HTx patients at scheduled biopsies (1 or 2 years after implantation)

Study 2: Development in cardiac and mitochondrial function following HTx Design: Mitochondrial function measured at scheduled EBM follow-up (1,2,3,4,8,12 weeks and 6 months after HTx) from 24 HTx patients. These results are compared to 15 patients with biopsies performed at 1 and 2 years after HTx.

Study 3: The impact of coronary arterial vasculopathy on mitochondrial function Design: Mitochondrial function assessed at scheduled EMB follow-up visits of patients with CAV as determined by coronary angiography (scheduled procedure) 15 HTx patients CAV are compared to 15 HTx patients with without CAV.

Study 4: MEE as a non-invasive marker of mitochondrial function and allograft rejection Design: 24 HTX patients scheduled for EMB will be examined twice with 11C-acetate-PET. It is intended that we consecutively recruit patients enrolled in study 2. The first examination is performed within 3 weeks following HTx and the second examination after 6 months. Up to 4 weeks between EMB and the second 11C-acetate PET examination is accepted.

(The HTx patient cohort which is subjected to biopsies 1 and 2 years after HTx in study 3 (n=15) is reused in study 1 and 2 as a comparable cohort. Hence, a total of 69 patients are enrolled. However, it is anticipated that several patients from study 1 and are enrolled in study 2 which will decrease the total number of participants.)

Methods

Mitochondrial function will be assessed in myocardial biopsies by High-resolution respirometry and Electron microscopy

Cardiac functions is assessed by transthoracic echocardiography

Coronary Angiography is performed to assess the degree of CAV

Blood samples will be taken

In study 4, MEE will be assessed by positron emission tomography using validated kinetic methods.

Ethical considerations

The project will be carried out in accordance with the principles of the Helsinki Declaration II. The protocol, including the written participant information and consent forms must be finally approved by the Research Ethics Committee of the Central Denmark Region and .

Publication and study plan All results, whether positive, negative or inconclusive will be published in an international peer-reviewed scientific journal.

Perspectives Cellular rejection (ACR) shortly after HTx is strongly associated with the long-term development of CAV and subsequent myocardial dysfunction. As graft failure and CAV are the major long-term heart-related late mortality causes following HTx, it seems paramount to modify long-term hazards such as ACR, CAV, and graft failure to significantly improve post-transplant outcome.5 In this context mitochondrial function seems to be pivotal, hence, approaches to assess mitochondrial function in HTx patient may prove to pave the way for new follow-up algorithms and even treatment targets.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent from participants

Exclusion Criteria:

* Under 18 years of age
* Endomyocardial biopsy not feasible assessed by surgeon
* Pregnancy (Study 4 only)
* Myocardial infarction, or hospitalization within 1 month due to any cardiac cause (Study 4 only)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: HTx patients Patients older than 18 years old can be included in this study provided that they give written consent. Pregnant women will not be included in study 4 because of a risk of genetic modifications based on the radiation from the PET-scans.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2019-04-25 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Study 1+3: Differences in Mitochondrial oxidative capacity | unpaired comparison differences between groups through study completion, an average of 2 years)
  Mitochondrial respiratory capacity evaluated with high resolution respirometry,
Study 2: Changes in mitochondrial oxidative capacity | unpaired comparison differences between groups (through study completion, an average of 2 years)
  Changes in mitochondrial respiratory capacity evaluated with high resolution respirometry,
Study 4: Changes in myocardial external energy efficiency | Changes from baseline (following HTX) to 6-month post-HTX (paired data)
  Changes Myocardial external energy efficiency evaluated by PET-scans with 11C-acetate tracer.
  Calculated by the ratio of myocardial external work (EW) and oxidative metabolism (MVO2).

SECONDARY OUTCOMES:
Biochemistry | Through study completion, an average of 2 years.
  TNT, proBNP, IL-1, IL-6, TNFalpha, sST2
Cardiac function | Through study completion, an average of 2 years.
  Left ventricular function (GLS) assessed by echocardiography
Invasive hemodynamics | Through study completion, an average of 2 years.
  Pulmonary (mPAP) and wedge pressures (mPCWP) assessed by right heart catheterization
Cellular function | Through study completion, an average of 2 years.
  Rejection state in cardiac tissue (assessed on the international scale for tissue rejection by pathologist):
  Grade 0R - No rejection. Grade 1R, mild - Interstitial and/or perivascular infiltrate with up to 1 focus of myocyte damage.
  Grade 2R, moderate - Two or more foci of infiltrate with associated myocyte damage.
  Grade 3R, severe Diffuse infiltrate with multifocal myocyte damage ± edema, ± hemorrhage ± vasculitis.
Mitochondrial structure | Through study completion, an average of 2 years.
  Assessed by electron microscopy (mitochondrial density and matrix folding)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Eiskjær, Prof., Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital Department of Cardiology, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clemmensen TS, Logstrup BB, Eiskjaer H, Poulsen SH. Serial changes in longitudinal graft function and implications of acute cellular graft rejections during the first year after heart transplantation. Eur Heart J Cardiovasc Imaging. 2016 Feb;17(2):184-93. doi: 10.1093/ehjci/jev133. Epub 2015 Jun 1. PMID 26034093
- [Background] Di Lisa F, Bernardi P. Mitochondria and ischemia-reperfusion injury of the heart: fixing a hole. Cardiovasc Res. 2006 May 1;70(2):191-9. doi: 10.1016/j.cardiores.2006.01.016. Epub 2006 Feb 23. PMID 16497286
- [Background] DePasquale EC, Ardehali A. Primary graft dysfunction in heart transplantation. Curr Opin Organ Transplant. 2018 Jun;23(3):286-294. doi: 10.1097/MOT.0000000000000523. PMID 29553954
- [Background] Sipahi I, Starling RC. Cardiac allograft vasculopathy: an update. Heart Fail Clin. 2007 Jan;3(1):87-95. doi: 10.1016/j.hfc.2007.02.007. PMID 17545012
- [Background] Lund LH, Edwards LB, Kucheryavaya AY, Benden C, Dipchand AI, Goldfarb S, Levvey BJ, Meiser B, Rossano JW, Yusen RD, Stehlik J. The Registry of the International Society for Heart and Lung Transplantation: Thirty-second Official Adult Heart Transplantation Report--2015; Focus Theme: Early Graft Failure. J Heart Lung Transplant. 2015 Oct;34(10):1244-54. doi: 10.1016/j.healun.2015.08.003. Epub 2015 Aug 28. No abstract available. PMID 26454738
- [Background] Kobayashi Y, Kobayashi Y, Yang HM, Bouajila S, Luikart H, Nishi T, Choi DH, Schnittger I, Valantine HA, Khush KK, Yeung ACY, Haddad F, Fearon WF. Long-term prognostic value of invasive and non-invasive measures early after heart transplantation. Int J Cardiol. 2018 Jun 1;260:31-35. doi: 10.1016/j.ijcard.2018.01.070. PMID 29622448
- [Background] Schneeberger S, Amberger A, Mandl J, Hautz T, Renz O, Obrist P, Meusburger H, Brandacher G, Mark W, Strobl D, Troppmair J, Pratschke J, Margreiter R, Kuznetsov AV. Cold ischemia contributes to the development of chronic rejection and mitochondrial injury after cardiac transplantation. Transpl Int. 2010 Dec;23(12):1282-92. doi: 10.1111/j.1432-2277.2010.01126.x. PMID 20561305
- [Background] Ventura-Clapier R, Garnier A, Veksler V. Energy metabolism in heart failure. J Physiol. 2004 Feb 15;555(Pt 1):1-13. doi: 10.1113/jphysiol.2003.055095. Epub 2003 Dec 5. PMID 14660709
- [Background] Gvozdjakova A, Kucharska J, Mizera S, Braunova Z, Schreinerova Z, Schramekova E, Pechan I, Fabian J. Coenzyme Q10 depletion and mitochondrial energy disturbances in rejection development in patients after heart transplantation. Biofactors. 1999;9(2-4):301-6. doi: 10.1002/biof.5520090227. PMID 10416044
- [Background] Gormsen LC, Svart M, Thomsen HH, Sondergaard E, Vendelbo MH, Christensen N, Tolbod LP, Harms HJ, Nielsen R, Wiggers H, Jessen N, Hansen J, Botker HE, Moller N. Ketone Body Infusion With 3-Hydroxybutyrate Reduces Myocardial Glucose Uptake and Increases Blood Flow in Humans: A Positron Emission Tomography Study. J Am Heart Assoc. 2017 Feb 27;6(3):e005066. doi: 10.1161/JAHA.116.005066. PMID 28242634
- [Background] Brown DA, Perry JB, Allen ME, Sabbah HN, Stauffer BL, Shaikh SR, Cleland JG, Colucci WS, Butler J, Voors AA, Anker SD, Pitt B, Pieske B, Filippatos G, Greene SJ, Gheorghiade M. Expert consensus document: Mitochondrial function as a therapeutic target in heart failure. Nat Rev Cardiol. 2017 Apr;14(4):238-250. doi: 10.1038/nrcardio.2016.203. Epub 2016 Dec 22. PMID 28004807
- [Background] Jespersen NR, Yokota T, Stottrup NB, Bergdahl A, Paelestik KB, Povlsen JA, Dela F, Botker HE. Pre-ischaemic mitochondrial substrate constraint by inhibition of malate-aspartate shuttle preserves mitochondrial function after ischaemia-reperfusion. J Physiol. 2017 Jun 15;595(12):3765-3780. doi: 10.1113/JP273408. Epub 2017 Feb 27. PMID 28093764
- [Background] Hansson NH, Harms HJ, Kim WY, Nielsen R, Tolbod LP, Frokiaer J, Bouchelouche K, Poulsen SH, Wiggers H, Parner ET, Sorensen J. Test-retest repeatability of myocardial oxidative metabolism and efficiency using standalone dynamic 11C-acetate PET and multimodality approaches in healthy controls. J Nucl Cardiol. 2018 Dec;25(6):1929-1936. doi: 10.1007/s12350-018-1302-z. Epub 2018 May 31. PMID 29855984
- [Background] Mehra MR, Crespo-Leiro MG, Dipchand A, Ensminger SM, Hiemann NE, Kobashigawa JA, Madsen J, Parameshwar J, Starling RC, Uber PA. International Society for Heart and Lung Transplantation working formulation of a standardized nomenclature for cardiac allograft vasculopathy-2010. J Heart Lung Transplant. 2010 Jul;29(7):717-27. doi: 10.1016/j.healun.2010.05.017. PMID 20620917